CLINICAL TRIAL: NCT06322251
Title: Identifying Intimate Partner Violence: an Intervention Study in Health Care Using a Standardised Questionnaire and Virtual Patients
Brief Title: Identification of Interpesonal Violence
Acronym: ViP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Linkoeping University (Other Government); Karolinska Institutet (Other); Stockholm University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-03399-01
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-01

CONDITIONS: Primary Health Care; Interpersonal Violence; Youth; Pregnancy
Keywords: Youth; Pregnancy; Primary care; Virtual patient; Interpersonal violence

STUDY DESIGN:
Intervention Model Description: Baseline measure - Number of patients that are identified fo being exposed to violence.
  Intervention:
  There are three settings:
  1. Primary Care Health Centers
  2. Youth Clinics
  3. Maternity Clinics
  At each type of clinic, the following interventions will be applied:
  Identification of domestic violence through
  1. Use of Virtual patient
  2. use of screening questionnaire
  3. a combination of a and b above.
  The clinics will randomised to either condition a, b or c.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Use of questionnaire (Other): Intervention I: Over a period of two months, healthcare professionals will ask standardized questions about exposure to violence using a questionnaire that measures exposure to physical, psychological, and sexual violence over the past 12 months. These questions will be verbally asked to all patients visiting the care units, regardless of the reason for their visit.
  Interventions: Behavioral: Use of instrument to identify exposure to violence in close relationships
- Use of virtual patient (Other): Intervention II: Healthcare professionals will undergo training to ask questions about violence in close relationships and practice how to utilize the answers, determine necessary care and interventions, and refer patients further. This training will utilize a "virtual patient" scenario where users interact with a realistic simulated patient through recorded video sequences. The training with the virtual patient will be conducted individually. On the digital platform, users will have access to the patient's medical background and other relevant information. Users can choose questions from a question bank, and based on their choices, they will receive feedback from both the patient and experts on their questions and treatment in the final part of the platform.
  Interventions: Behavioral: Use of instrument to identify exposure to violence in close relationships
- Combined use of questionnaire and virtual patient (Other): Intervention III: This intervention combines Intervention I and II methods. Participants will investigate the identification of intimate partner violence over a two-month period after training with the virtual patient and in parallel with administering the violence questionnaire.
  Interventions: Behavioral: Use of instrument to identify exposure to violence in close relationships

INTERVENTIONS:
Behavioral: Use of instrument to identify exposure to violence in close relationships — Use of instrument to identify exposure to violence in close relationships
  Other Names: Use of Questionnaire; Use of Virtual patient; Use of a combination of questionnaire and virtual patient

SUMMARY:
The goal of this study is to increase primary care professional's ability to identify individuals exposed to intimate partner violence (IPV) in primary health care settings.

The main questions it aims to answer are

1. To what extent do the following three interventions contribute to identify potential victims of IPV: (1) the use of a standardized questionnaire that screens exposure to IPV, (2) staff using tailored virtual patients for clinical training on IPV and (3) a combination of interventions 1 and 2?
2. Which intervention do primary care professionals experience as most effective in increasing the ability to identify and respond to victims of IPV?

Participants will be divided to apply one of the three interventions in their health care setting: 1) a standardized questionnaire to patients, 2) virtual patients tailored to health professionals, and 3) a combination of 1 and 2.

Pre-and post-measurement of the health professionals identification of patients exposed to IPV will will be used to explore the effect of the interventions.

Focus group interviews with the participating health professionals will be a qualitative complement. The participants will be asked about what intervention they experience as the most effective in increasing the ability to identify victims of IPV.

DETAILED DESCRIPTION:
The project is expected to last for three years and is based on a quasi-experimental design. The outcome is the registration of the number of individuals exposed to intimate partner violence, which will be investigated before and after intervention. Qualitative focus group interviews with participating healthcare professionals will also be included to investigate which intervention they perceive as most effective in increasing the ability to identify people exposed to intimate partner violence. The project will be carried out at different care units in primary care (health centers, midwifery clinics, youth clinics), and healthcare professionals will be randomized based on the following three interventions:

1. Use of a standardized questionnaire.
2. Training in asking questions about intimate partner violence via training with tailored virtual patients.
3. A combination of interventions 1 and 2.

To measure the outcome of the project, the research group will use registry data (health centers/youth clinics) and a protocol (midwifery clinics) to record the number of patients exposed to intimate partner violence.

The research subjects in this project are primarily participating healthcare professionals involved in the interventions. The nature of data from the research subjects primarily consists of background information such as demographic data (e.g., age, level of education, occupational category, gender, professional experience), and whether healthcare professionals have undergone any training on IPV. This data should not be used in any analyses but only constitutes a descriptive description of the research subjects when data will be presented in scientific papers. Qualitative focus group interviews with participating healthcare professionals will also be included to investigate which intervention they experience as most effective in increasing the ability to identify people exposed to intimate partner violence.

Registry data for patients who have visited health centers and youth clinics will be collected retrospectively from the Center for Health Data in Region Stockholm. Sociodemographic information about visitors to health centers and youth clinics is obtained from Statistics Sweden's population register; however, names and social security numbers are not conveyed to the research group. Pseudonymization is carried out, and the code key is stored at the Centre for Health Data. In the protocols, midwifery clinics will note the number of patients who state exposure to violence in close relationships, reasons for seeking treatment, support measures taken by healthcare staff, and whether the patient is exposed to violence.

Data will be measured at the group level within participating activities. Validity may become uncertain if healthcare professionals forget to document information in medical records or protocols, or if there are healthcare professionals who do not want to participate in the intervention. To counteract this, each participating unit will have a contact person who will be available and in regular contact with the unit. Before the intervention starts, members of the research team will also provide information about the study and approach.

Regarding the qualitative design, reliability is of paramount importance. Therefore, we will thoroughly describe data collection and the process of data analysis.

The analysis will primarily involve pre- and post-measurements of the interventions. Additionally, the reseachers will employ statistical analyses to compare the identification of cases of intimate partner violence among the three different interventions (comparisons between intervention groups). The researches will investigate whether the number of patients registered as victims of intimate partner violence has increased at each care unit after participants have undergone the study's interventions. Measurements will be conducted at the group level based on the participating care units, with the analysis focusing primarily on pre- and post-measurements.

Furthermore, the researchers will compare whether the number of registered cases of intimate partner violence differs between the three different interventions (comparison between intervention groups). This will be analyzed through regression analyses, where pre- and post-measurement is included as an interaction variable (time-after) x group (intervention).

The focus group interviews will be recorded, transcribed, and analyzed using inductive thematic analysis. Inductive analysis involves encoding data without attempting to fit it into a pre-existing coding template or the researcher's analytical starting points. This approach ensures that the thematic analysis remains data-driven.

ELIGIBILITY:
Inclusion criteria:

* All health care staff who meet patients at the included study sites are elegible for the study
* Midwives, MDs, psychologists, social workers, nurses etc.

Exclusion criteria:

- Health care staff who does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of identified persons seeking healthcare who have been exposed to violence | Baseline
  Comparison between before and after intervention - Effectiveness within intervention

SECONDARY OUTCOMES:
Number of identified persons seeking healthcae who have been exposed to violence | After the intervention during a period of 2 months
  Comparison between different interventions (Effectiveness between interventions)

OTHER OUTCOMES:
Experiences of health care staff | Three months after the intervention
  Experiences of health care staff to use questionnaire / virtual patient will be obtained in interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Mia M Barimani, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No